CLINICAL TRIAL: NCT02984293
Title: Impact of LILRB5 Genotype on Immune Response to Atorvastatin
Brief Title: Statin Immune Study
Acronym: ImmunoStat
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: NHS Tayside (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2016CV05; 16/ES/0128 (Other: East of Scotland Research Ethics Service)
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Last update posted 2018-12-03 (Actual); Status verified 2018-03

CONDITIONS: Drug Intolerance
Keywords: Atorvastatin; LILRB5; Statin intolerance
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atorvastatin (Active Comparator): The participants will receive atorvastatin (80 mg) orally once daily for 28 days.
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator): The participants will receive matched placebo orally once daily for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 80 mg once daily for 28 days.
  Arms: Atorvastatin
Drug: Placebo — Placebo once daily for 28 days.
  Arms: Placebo

SUMMARY:
Statins are widely used drugs to treat hypercholesterolaemia. In general, they are very safe drugs. However, up to one third of statin users can experience muscle symptoms, which are most commonly mild without any conventional laboratory signs of muscle damage. However, these muscle symptoms can often lead to poor compliance to the cholesterol-lowering therapy, reducing its effectiveness. Recent data has highlighted the potential role of immune system in development of statin-induced muscle pain. Variation in the LILRB5 gene has been associated with statin intolerance. We aim to investigate the impact of LILRB5 genetic variability in tolerability and immune response to atorvastatin in healthy volunteers.

The study is being undertaken at the Tayside Institute for Cardiovascular Research (TICR) in Ninewells Hospital, Dundee. We will recruit participants who have donated a sample to GoSHARE study. The participants will be healthy, and recruited according to their genotype of LILRB5 (information available from GoSHARE). The volunteers will then enter a randomised cross-over study with two treatment periods. During treatment period one, all participants will be commenced on atorvastatin or placebo (a dummy drug). Before and at the end of the treatment period, blood and urine samples will be taken and a muscle symptoms questionnaire will be completed to assess the tolerability and immune response to the study drug exposure. After four weeks, the study drug is stopped for a washout period of three weeks before cross-over commences. Thereafter, during treatment period two, the alternate study drug will be started, and tolerability will be assessed similar to that in period one. The study will last approximately 11 weeks. The volunteers have a total of 5 visits to the TICR.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-69 years
* Statin-naïve
* White European
* Healthy
* Acceptable laboratory test results

Exclusion Criteria:

* Significant disease
* Regular drug therapy
* Recent involvement (<30 days) in a CTIMP
* Inability/unwillingness to comply with the protocol
* Carry the rare variant of the CKM polymorphism rs11559024
* Unable to consent
* Woman of childbearing potential (i.e. premenopausal female capable of becoming pregnant)

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2017-11-03 (Actual); Study Completion 2017-11-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the change in CK levels at the end of the treatment from baseline in both treatment periods. | Measured at baseline (day 0) and day 29 of both treatment periods.

CONTACTS AND LOCATIONS:
Overall Officials: Colin NA Palmer, PhD FSB FRSE, Study Chair — University of Dundee
Locations (1):
- University of Dundee, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
As per GoSHARE tissue bank protocol, the data derived from the existing samples will be returned to the tissue bank for research use.

REFERENCES:
- [Background] Dube MP, Zetler R, Barhdadi A, Brown AM, Mongrain I, Normand V, Laplante N, Asselin G, Zada YF, Provost S, Bergeron J, Kouz S, Dufour R, Diaz A, de Denus S, Turgeon J, Rheaume E, Phillips MS, Tardif JC. CKM and LILRB5 are associated with serum levels of creatine kinase. Circ Cardiovasc Genet. 2014 Dec;7(6):880-6. doi: 10.1161/CIRCGENETICS.113.000395. Epub 2014 Sep 11. PMID 25214527
- [Background] Alfirevic A, Neely D, Armitage J, Chinoy H, Cooper RG, Laaksonen R, Carr DF, Bloch KM, Fahy J, Hanson A, Yue QY, Wadelius M, Maitland-van Der Zee AH, Voora D, Psaty BM, Palmer CN, Pirmohamed M. Phenotype standardization for statin-induced myotoxicity. Clin Pharmacol Ther. 2014 Oct;96(4):470-6. doi: 10.1038/clpt.2014.121. Epub 2014 Jun 4. PMID 24897241